CLINICAL TRIAL: NCT02759900
Title: Using a Cold Atmospheric Plasma Device to Treat Skin Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Skin Center Dermatology Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130084
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Actinic Keratosis; Acne/Rosacea; Verruca Plana; Tinea; Molluscum Contagiosum; Bowen's Disease; Warts
MeSH Terms: conditions — Keratosis, Actinic; Rosacea; Tinea; Molluscum Contagiosum; Bowen's Disease; Warts

ARMS (2):
- Non-thermal atmospheric plasma treatment (Experimental): Device treatment
  Interventions: Device: Non-thermal, atmospheric plasma to treat skin lesions and acne
- Indirect non-thermal atmospheric plasma treatment (Experimental): A compound of non-thermal atmospheric plasma and medium is used to treat the target by direct application or by on-site generation of the compound
  Interventions: Device: Indirect non-thermal, atmospheric plasma to treat hair loss and acne

INTERVENTIONS:
Device: Non-thermal, atmospheric plasma to treat skin lesions and acne — Non-thermal, atmospheric plasma treatment of affected area or lesions using a nanosecond dielectric barrier discharge plasma device
  Arms: Non-thermal atmospheric plasma treatment
Device: Indirect non-thermal, atmospheric plasma to treat hair loss and acne — A compound of non-thermal, atmospheric plasma and medium is delivered to or generated at the target area. Plasma is generated using either microsecond dielectric barrier discharge plasma device or PiezoBrush (a helium jet plasma). The medium is an aqueous alcohol solution
  Arms: Indirect non-thermal atmospheric plasma treatment

SUMMARY:
This study examines the efficacy of a non-thermal, atmospheric plasma device in the treatment of skin disorders

DETAILED DESCRIPTION:
The study uses non-thermal atmospheric pressure plasma to treat target conditions. The patients are monitored at set intervals for efficacy and adverse effects using investigator's assessment and imaging techniques

ELIGIBILITY:
Inclusion Criteria:

* diagnoses of target conditions
* ability to complete study protocol

Exclusion Criteria:

* based on specific condition

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 1-12 months
  The outcome is the presence or lack of clinical improvement in the investigator's global assessment and reviewing photo-documentation as well as reflectance confocal microscopy study investigator's global assessment and reviewing photo-documentation

CONTACTS AND LOCATIONS:
Locations (1):
- The Skin Center Dermatology Group, New City, New York, United States

REFERENCES:
- [Derived] Friedman PC, Fridman G, Fridman A. Cold atmospheric pressure plasma clears molluscum contagiosum. Exp Dermatol. 2023 Apr;32(4):562-563. doi: 10.1111/exd.14695. Epub 2022 Nov 3. No abstract available. PMID 36302167
- [Derived] Malik S, Gill M, Fridman G, Fridman A, Friedman PC. Cold atmospheric plasma reduces demodex count on the face comparably to topical ivermectin, as measured by reflectance confocal microscopy. Exp Dermatol. 2022 Sep;31(9):1352-1354. doi: 10.1111/exd.14584. Epub 2022 May 11. No abstract available. PMID 35491738